CLINICAL TRIAL: NCT05347797
Title: Phase 3 Multicentre, Prospective, Interventional Clinical Study Testing DNA Extracted From Tumour Tissue Biopsy Samples, Using the Therascreen® KRAS RGQ PCR Kit, From Patients With Non-Small Cell Lung Cancer, Screened in Clinical Study (Protocol No. 20190009).
Brief Title: Clinical Study Testing DNA Extracted From Tumour Tissue Biopsy Samples, Using the Therascreen® KRAS RGQ PCR Kit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: QIAGEN Gaithersburg, Inc (Industry)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: QMAN-18-0181-1-003
Record Dates: First submitted 2022-04-01; First posted 2022-04-26 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Clinical Performance Study Protocol for therascreen® KRAS RGQ PCR Kit (Other): The KRAS Kit is a real-time qualitative PCR assay used on the Rotor-Gene Q MDx instrument for the detection of somatic G12C mutations in the human KRAS oncogene using DNA extracted from formalin fixed paraffin-embedded (FFPE) Non-small Cell Lung Cancer (NSCLC) tissue. The KRAS Kit is intended to aid in the identification of cancer patients who may be eligible for treatment with AMG 510.
  Interventions: Diagnostic Test: therascreen® KRAS RGQ PCR Kit

INTERVENTIONS:
Diagnostic Test: therascreen® KRAS RGQ PCR Kit — To utilize a Clinical Study assay, the therascreen® KRAS RGQ PCR Kit, as a screening test in Phase 3 of Clinical Study (Protocol No. 20190009), in order to identify patients with NSCLC with KRAS G12C mutation positive tumours.

SUMMARY:
An interventional, prospective study. It is estimated that up to 800 patient tissue samples (from approximately 650 patients enrolled at approximately 300 clinical trial sites), will be obtained as part of enrolment into Phase 3 of Clinical Study (Protocol No. 20190009), for testing using the therascreen® KRAS RGQ PCR Kit (KRAS Kit).

DETAILED DESCRIPTION:
This is an interventional, prospective clinical performance study protocol, for the testing of DNA extracted from tumour tissue biopsy samples (resected and core needle biopsy [CNB]/fine needle aspiration [FNA]) tumour tissue ) obtained from patients with Non-Small Cell Lung Cancer (NSCLC), using the KRAS Kit.

Up to 800 patient tissue samples (from approximately 300 clinical trial sites), obtained in the Clinical Study (Protocol No. 20190009), will be tested using the KRAS Kit. The testing will be performed at the investigational device clinical testing sites, Q2 Solutions Laboratories in the four geographical locations: USA, Singapore, UK and China.

The primary objective of the Clinical Study (Protocol No. 20190009) is to evaluate tumour objective response rate (ORR) assessed by MODIFIED RECIST 1.1 criteria of AMG 510 as a monotherapy in patients using the Clinical Study Assay, KRAS Kit to assess whether to treat patients with KRAS G12Cmutated advanced tumours (NSCLC).

The clinical data from the study will be used to determine the drug-device efficacy to support future regulatory submissions for the device-drug combination.

ELIGIBILITY:
Inclusion Criteria:

* All patients who provided consent (by signing and dating the ICF for Protocol No. 20190009), may be included in the Clinical Performance Study.

Exclusion Criteria:

* Patients whose tumour tissue biopsy samples are not Clinical Study Assay evaluable will be asked to provide further tumour tissue biopsy samples. Patients with samples identified for the study which have insufficient testing material will have their sample excluded, as will specimens which have undergone decalcification.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 495 (Actual)
Dates: Start 2020-03-13 (Actual); Primary Completion 2021-04-22 (Actual); Study Completion 2021-04-22 (Actual)

PRIMARY OUTCOMES:
therascreen® KRAS RGQ PCR Kit (KRAS Kit). | 5 business days
  To utilize the Clinical Trial Assay, the (KRAS Kit), as a screening test in Phase 3 of Clinical Study (Protocol No. 20190009), in order to identify patients with NSCLC who have the KRAS G12C mutation.

CONTACTS AND LOCATIONS:
Locations (1):
- QIAGEN Gaithersburg, Inc, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No